CLINICAL TRIAL: NCT02155946
Title: Promoting Adaptive Neuroplasticity in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N1534-R
Record Dates: First submitted 2014-05-29; First posted 2014-06-04 (Estimated); Results first posted 2022-09-01 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Aging; Alzheimer's Disease/Dementia; Cognitive Disorders; Imaging; Magnetic Resonance Imaging (MRI); Neurology; Physical Medicine & Rehabilitation; transcranial direct current stimulation
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- active tDCS + mnemonic strategy training (Experimental): Group receives active brain stimulation plus memory rehabilitation
  Interventions: Device: Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit
- sham tDCS + mnemonic strategy training (Active Comparator): Group receives sham brain stimulation plus memory rehabilitation
  Interventions: Device: Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit
- active tDCS + autobiographical memory recall (Active Comparator): Group receives active brain stimulation plus reminiscence training
  Interventions: Device: Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit
- sham tDCS + autobiographical memory recall (Active Comparator): Group receives sham brain stimulation plus reminiscence training
  Interventions: Device: Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit — Active brain stimulation
  Arms: active tDCS + autobiographical memory recall; active tDCS + mnemonic strategy training
Device: Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit — Sham (placebo)
  Arms: sham tDCS + autobiographical memory recall; sham tDCS + mnemonic strategy training

SUMMARY:
The aging US population threatens to overwhelm our healthcare infrastructure, especially since the rate of Alzheimer's disease (AD) alone is expected to triple in the coming decades. Memory cause functional impairment, reduced quality of life, increased caregiver burnout, and eventual institutionalization. The diagnosis of mild cognitive impairment (MCI) identifies those with memory deficits but who remain relatively independent in everyday life. MCI provides a window for interventions that target memory functioning. The proposed study focuses specifically on a groundbreaking combination of mnemonic rehabilitation and non-invasive brain stimulation. The main idea is that brain stimulation can enhance functioning in the specific brain regions/networks, thereby increasing the patients' ability to benefit from different types of memory rehabilitation. This will be a randomized, double-blind study (active vs. fake brain stimulation), that provides multiple treatment session. Outcome will be examined using both laboratory-based and real-world memory testing as well as brain imaging. This first-of-its-kind study has the potential to meaningfully translate more "basic" science findings into neuroanatomically targeted and functionally meaningful treatments for our aging population.

DETAILED DESCRIPTION:
Enrollment and interactions/interventions are temporarily paused due to COVID-19 and are expected to resume in the future. This is not a suspension of IRB approval.

The proposed study focuses specifically on a groundbreaking combination of mnemonic rehabilitation and non-invasive brain stimulation. The main idea is that brain stimulation can enhance functioning in the specific brain regions/networks, thereby increasing the patients' ability to benefit from memory rehabilitation. This will be a randomized, double-blind study (active vs. fake brain stimulation), that provides multiple treatment session. Outcome will be examined using both laboratory-based and real-world memory testing as well as brain imaging. This first-of-its-kind study has the potential to meaningfully translate more "basic" science findings into neuroanatomically targeted and functionally meaningful treatments for our aging population.

The general purpose of this study is to examine the effects of two types of treatments for memory impairment in those with mild cognitive impairment (MCI). One form of treatment is cognitive rehabilitation, which involves teaching new ways to learn and remember information. The second form of treatment uses a type of electrical brain stimulation called transcranial direct current stimulation (tDCS) to increase activity in certain brain areas that may be involved with memory. We will use brain imaging to see whether these treatments changed how individuals learn and remember information. We will also use cognitive tests and questionnaires to examine whether memory (and related abilities) changed because of treatment.

Values were updated in February 2023 after discovering coding errors in the original database. An exploratory outcome variable (effect of brain volumes) was removed at that time since the electrical field analyses are fundamentally dependent on brain volumes - the EF outcome measure remained but was modified to remove the two sham conditions since, by design, they did not receive any electric field (i.e., sham) and the statistical corrections could not be performed.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria (all patients):

* All medications stable for approximately 2-3 months;
* No history of severe mental illness;
* No current untreated alcohol or substance abuse/dependence;
* English as native and preferred language;
* MRI-compatible if taking part in fMRI studies
* Able to give informed consent.

MCI Inclusion Criteria:

- Diagnosis of amnestic MCI based on criteria set forth by Petersen (2004). Additionally, other potential causes of cognitive deficit ruled out by the referring physician

Exclusion Criteria:

* History of neurological disease or injury
* History of severe mental illness
* Current untreated alcohol or substance abuse
* Other conditions may exclude; please discuss with contact

Ages: 50 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M. Hampstead, PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Group receives active brain stimulation plus mnemonic strategy training
  Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit: Active brain stimulation
- Arm 2: Group receives sham brain stimulation plus mnemonic strategy training
  Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit: Sham (placebo)
- Arm 3: Group receives active brain stimulation plus autobiographical recall
  Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit: Active brain stimulation
- Arm 4: Group receives sham brain stimulation plus autobiographical recall
  Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit: Sham (placebo)
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 29 | 25 | 29 | 24
Completed | 29 (number completed at primary endpoint) | 23 (number completed at primary endpoint) | 29 (number completed at primary endpoint) | 24 (number completed at primary endpoint)
Not Completed | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 3: Group receives active brain stimulation plus autobiographical memory recall
  Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit: Active brain stimulation
- Arm 4: Group receives sham brain stimulation plus autobiographical memory recall
  Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit: Sham (placebo)
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 29 | 25 | 29 | 24 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.59 (7.31) | 73.88 (6.08) | 72.31 (7.36) | 74.04 (6.2) | 73.14 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 11 | 12 | 42
  Male | 16 | 19 | 18 | 12 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 3 | 1 | 11
  White | 24 | 23 | 26 | 23 | 96
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 25 | 29 | 24 | 107

OUTCOME MEASURES:

1. Primary Outcome: Face-name Memory Test Performance
Description: Raw number of face-name pairs correctly recalled with a maximum of 15 points; higher values are better at each time point. Change at post-session 5 (day 5 after baseline)) calculated relative to baseline performance (positive differences indicate improvement; negative values indicate decline). Data coding errors were identified and accurate values were reported 2/6/2023.
Time Frame: change from baseline to post session 5 (day 5 after baseline)
Population: Patient-level factors of age, sex, race, RBANS Delayed Memory Index, MoCA, Emory version of the Wisconsin Card Sorting Test were included as covariates.
Measure: Mean (95% Confidence Interval); unit: pairs correctly recalled/recognized
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 29 | 23 | 29 | 24
pairs correctly recalled/recognized | -.28 [-1.29 to .74] | -.01 [-1.15 to 1.13] | -1.29 [-2.33 to -.24] | -1.76 [-2.86 to -.66]

2. Primary Outcome: Object Location Association Memory Test Performance - Recognition Condition
Description: Performance measured using number of correctly identified locations (3 locations per stimulus; 15 total stimuli). Higher values indicate better performance. Change at post-session 5 (day 5 after baseline) calculated relative to baseline performance (positive differences indicate improvement; negative values indicate decline). Data coding errors were identified and accurate data were updated 2/6/2023.
Time Frame: change from baseline to post session 5 (day 5 after baseline)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Number correct relative to baseline
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 29 | 23 | 29 | 24
Number correct relative to baseline | .55 [-.48 to 1.58] | .25 [-.9 to 1.4] | .07 [-.98 to 1.12] | -.76 [-1.87 to .35]

3. Primary Outcome: fMRI Betaweight Change
Description: Changes in task related blood oxygen dependent signal (BOLD) activation for the face-name (novel post > novel pre) contrast in the left inferior frontal gyrus (pars triangularis, pars orbitalis, pars opercularis). Data are preliminary betaweights for the above noted contrast. Positive values reflect increased BOLD signal while negative values represent reduced BOLD signal. Not all participants were able to complete fMRI, which explains sample size discrepancies with other outcome measures. Data coding errors were discovered and accurate, updated data reported on 2/6/2023
Time Frame: change from baseline to post session 5 (day 5 after baseline)
Measure: Mean (95% Confidence Interval); unit: Percent BOLD signal change
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 23 | 21 | 20 | 20
Percent BOLD signal change | .34 [.08 to .59] | -.09 [-.36 to .18] | .07 [-.22 to .35] | -.13 [-.39 to .13]

4. Secondary Outcome: Prose Memory
Description: Performance on the Ecological Memory Simulations- Medical Instructions subtest. Raw points where higher values reflect better performance at each time point (0-15 possible points at each time point). Reported values reflect change from baseline (i.e., post-session day 5 vs. baseline) where positive values represent improvement and negative values represent decline. Corrected values are now included (2/23) that account for age, sex, and baseline neuropsychological abilities.
Time Frame: change from baseline to post Session 5 (day 5 after baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 29 | 23 | 29 | 24
units on a scale | -1.07 [-2.23 to .1] | -1.18 [-2.46 to .11] | -.93 [-2.13 to .26] | -1.56 [-2.81 to -.31]

5. Secondary Outcome: MMQ - Strategy Subscale
Description: Changes on the Multifactorial Memory Questionnaire - strategy subscale. Raw points where higher values reflect better performance at each time point (0-76 possible points at each time point). Reported values reflect change from baseline (i.e., post-session day 5 vs. baseline) where positive values represent improvement and negative values represent decline.
Time Frame: change from baseline to post session 5 (day 5 after baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 29 | 23 | 29 | 24
units on a scale | 1.41 [-.97 to 3.8] | 1.1 [-1.6 to 3.81] | -1.9 [-4.28 to .48] | -.5 [-3.12 to 2.12]

6. Secondary Outcome: Spatial Navigation
Description: Performance on Ecological Memory Simulations routes subtest (serial order). Higher values indicate better performance at each time point (0-9 possible points at each time point). Change from baseline is reported (post-session day 5 vs. baseline) so higher values indicate better recall while negative values indicate decline. Corrected data are now reported (2/23) accounting for age, sex, and baseline neuropsychological abilities.
Time Frame: change from baseline to post session 5 (day 5 after baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 29 | 23 | 29 | 24
units on a scale | .59 [-.15 to 1.32] | .74 [-.08 to 1.55] | 1.03 [.27 to 1.79] | .6 [-.19 to 1.39]

7. Other Pre Specified Outcome: Planned (Tertiary) Analyses of Patient-specific Characteristics That Affect Treatment Outcome
Description: Planned analyses to examine patient specific characteristics that affect treatment efficacy and would be vital for clinical translation at the individual patient level. Data analyzed using a composite "recognition" score that combined the face-name and object-location task recognition scores (total on a 0-30 point scale; values below are change from baseline; higher values are "better" and reflect improved memory test performance). Patient-level factors of age, sex, race, RBANS Delayed Memory Index, MoCA, Emory version of the Wisconsin Card Sorting Test (total sorts) were included as covariates.
Time Frame: change from baseline post treatment (within ~ 96 hours of session 5)
Population: linear mixed model Data analyzed using a composite "recognition" total score that combined the face-name and object-location task (change on 0-30 point scale relative to baseline) higher scores are better). Patient-level factors of age, sex, race, RBANS Delayed Memory Index, MoCA, Emory version of the Wisconsin Card Sorting Test (total sorts) were included as covariates.
Measure: Mean (95% Confidence Interval); unit: change in total score on 30 point scale
Groups:
- Active tDCS + Autobiographical Memory Recall: Group receives active brain stimulation plus ABR
  Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit: Active brain stimulation
- Sham tDCS + Autobiographical Memory Recall: Group receives sham brain stimulation plus ABR
  Transcranial direct current stimulation (tDCS) Soterix Medical Inc. tDCS unit: Sham (placebo)
Arm/Group | Active tDCS + Mnemonic Strategy Training | Sham tDCS + Mnemonic Strategy Training | Active tDCS + Autobiographical Memory Recall | Sham tDCS + Autobiographical Memory Recall
Number analyzed (Participants) | 29 | 23 | 29 | 24
change in total score on 30 point scale | .28 [-1.23 to 1.79] | .09 [-1.62 to 1.79] | -1.12 [-2.68 to .43] | -2.52 [-4.15 to -.89]

8. Other Pre Specified Outcome: Change in Beta-weights Controlling for Electric Field (EF)
Description: Outcome measure is the change in betaweight (as a percent signal change: post session 5 minus baseline) during the face-name and object-location tasks (same metric as Primary Outcome measure 3) while controlling for the electric field (EF). Finite element model based measurement of electric field in the targeted brain regions (Values range from 0 to no theoretical upper limit with higher values reflecting more electrical current; most values will be under 0.5 V/m). The EF was calculated using the baseline MRI T1 scan for each individual. EF values were then included in the linear mixed model analysis of fMRI Beta-weight change (post training vs. baseline) since EF values at the targeted brain region varied across participants. Note, EF values only apply to active HD-tDCS groups, so sham groups have no data to report and were removed accordingly (updated 2/23).
Time Frame: Betaweight change: Post session 5 (day 5) minus baseline
Population: linear mixed model that includes EF as a predictor variable as well as covariates of age, sex, education, and race.
Measure: Mean (95% Confidence Interval); unit: % signal change (session 5 vs baseline)
Arm/Group | Active tDCS + Mnemonic Strategy Training | Active tDCS + Autobiographical Memory Recall
Number analyzed (Participants) | 23 | 20
% signal change (session 5 vs baseline) | .11 [-.08 to .3] | -.03 [-.22 to .16]

ADVERSE EVENTS:
Time Frame: Primary study intervention period (5 days)
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/23 | 0/29 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/23 | 0/29 | 0/24
Other Adverse Events (participants affected / at risk) | 0/29 | 0/23 | 0/29 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT02155946/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT02155946/SAP_001.pdf
  • Informed Consent Form (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT02155946/ICF_002.pdf